CLINICAL TRIAL: NCT04341064
Title: A Personalized Approach to Skin Cancer Prevention Among Adolescents
Brief Title: Sun-safe Habits Intervention and Education
Acronym: SHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yelena Wu, Assistant Professor, Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00118620; 1R01CA244674-01 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Skin Cancer; Adolescents
Keywords: Education; Prevention and Control; Behavioral Research
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHINE (Experimental): Participants will be randomized to receive an intervention that provides information on skin cancer and preventive strategies, features a personalized skin cancer prevention packet that focuses on students' UVR exposure and skin cancer risk, and includes the creation of a individualized sun protection action plan.
  Interventions: Behavioral: SHINE Intervention
- Standard Education (No Intervention): Participants will be randomized to receive information that covers general skin cancer education for pediatric populations.

INTERVENTIONS:
Behavioral: SHINE Intervention — [see arm/group descriptions]
  Arms: SHINE

SUMMARY:
The purpose of this study is to determine the efficacy of the Sun-safe Habits Intervention and Education (SHINE) intervention in improving sun protection use and decreasing intentional tanning among high school students. It's anticipated that 30 schools will be randomized into the trial, with approximately half assigned to SHINE and the other half assigned to standard education. After randomization and a baseline assessment, each school will receive two in-class intervention sessions delivered by an interventionist. Follow-up assessments will be completed one month post-intervention, 3-4 months post-intervention, one year post-baseline, and one year post-intervention.

DETAILED DESCRIPTION:
Enrollment: Recruitment will occur through schools and districts that are committed to partnering with the study team. Schools will be stratified into 2 groups and then randomized to receive either the SHINE intervention or standard education. Stratification will be based on school demographic factors. The investigators anticipate enrolling a total of 30 schools into the trial, with approximately half of schools assigned to the SHINE intervention. Prior to student enrollment, parents will be sent a cover letter describing the study and will be given the choice of opting their child out of the study. Students will receive an assent cover letter and will be given the choice of opting out of the study. With the exception of students who opt out of participation or are opted out by their parents, all students between the ages of 11 and 21 years present in class during the days of intervention delivery and assessments will receive the intervention and be asked to complete the assessments.

Intervention: After randomization, each school will receive the intervention materials for the condition to which they were assigned. Both SHINE and standard education groups will receive 2 in-class intervention sessions, each lasting 40 minutes each, and a 40-minute in-class booster sessions. Schools allocated to SHINE will create individualized action plans and receive personalized UV photos. Schools allocated to standard education will receive presentations of basic skin cancer prevention information available through the American Academy of Dermatology and Centers for Disease Control and Prevention.

Study Assessments: Regardless of which intervention group students are randomized to, they will be asked to complete 5 assessments. The first assessment (baseline) will occur in the fall. The intervention will be delivered in the spring. Approximately one month post-intervention, students will be asked to complete the first post-intervention assessment, followed by a summer assessment delivered 3-4 months post-intervention. Students will also be asked to complete two longer-term follow-up assessments at one year post-baseline and one-year post-intervention. All assessments will be completed via the web using REDCap. Each of these assessments is expected to take no more than 20 minutes. Students will be asked to provide information via questionnaire on sun protection behaviors, tanning behaviors, sunburn occurrence, self-efficacy and response efficacy related to skin cancer, susceptibility to skin cancer, severity of skin cancer, demographic characteristics, recall of the intervention, and knowledge and awareness of skin cancer prevention and risk.

ELIGIBILITY:
Inclusion Criteria:

Students are eligible for this trial if they:

* Attend high school in Utah (e.g. are enrolled in grades 9-12).

Exclusion Criteria:

Students will be excluded from participation if they:

* Do not speak English.
* Are unable to participant due to a developmental delay.

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2223 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Sunscreen Application Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in sunscreen application occurrence between timepoints.
  "These next questions ask about what you have typically done in the past month when you were outdoors in the sun for 1 hour or more. How often did you wear sunscreen?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Sunscreen Re-Application Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in sunscreen re-application occurrence between timepoints.
  "These next questions ask about what you have typically done in the past month when you were outdoors in the sun for 1 hour or more. How often did you re-apply sunscreen after being outside for 2 hours, in the water, or sweating?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Long Sleeved Shirt Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in long sleeved shirt occurrence between timepoints.
  "These next questions ask about what you have typically done in the past month when you were outdoors in the sun for 1 hour or more. How often did you wear a shirt with sleeves that covered your shoulders?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Long Pants/Skirt Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in long pants/skirt occurrence between timepoints.
  "These next questions ask about what you have typically done in the past month when you were outdoors in the sun for 1 hour or more. How often did you wear long pants or a long skirt?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Shade Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in shade occurrence between timepoints.
  "These next questions ask about what you have typically done in the past month when you were outdoors in the sun for 1 hour or more. How often did you stay in the shade or under an umbrella?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Peak Hours Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in avoidance of peak hours between timepoints.
  "These next questions ask about what you have typically done in the past month when you were outdoors in the sun for 1 hour or more. How often did you avoid being in the sun between 10:00AM-4:00PM?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Sunglasses Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in wearing sunglasses between timepoints.
  "These next questions ask about what you have typically done in the past month when you were outdoors in the sun for 1 hour or more. How often did you wear sunglasses?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Time Spent in the Sun to get Tan Behavior Changes Assessed Via Sun Habits Survey | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in time spent in the sun to get tan between timepoints.
  "These next questions ask about what you have done in the past (time frame) if you were outdoors in the sun for 15 minutes or more. How often did you spend time in the sun in order to get a tan?" Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Change in Tanning Behaviors Assessed Via Youth Risk Behavioral Surveillance System | Baseline Assessment (Wk 0), Post-Assessment (Wk 32-36), Follow-up #1 (Wk 36-40), Follow-up #2 (Wk 44-52), Follow-up #3 (Wk 84-88)
  Mean/standard deviation of the difference in student's indoor and outdoor tanning behaviors within the last month will be assessed using items from the Youth Risk Behavioral Surveillance System. Unintentional outdoor tanning will also be assessed.
  "In the past (time frame), how many times did you use an indoor tanning device such as a sunlamp, sunbed or tanning booth? (Do not count getting a spray-on tan)." Minimum value = 0; Maximum value = 5; Higher scores indicate a worse outcome
  "In the past (time frame), how many times did you sunbathe or tan outdoors?" Minimum value = 0; Maximum value = 5; Higher scores indicate a worse outcome
  "In the past (time frame), how many times did you end up with a tan, even if you didn't try to get one?" Minimum value = 0; Maximum value = 5; Higher scores indicate a worse outcome

SECONDARY OUTCOMES:
Change in Sunburn Occurrence Assessed Via Sun Habits Survey | Baseline (Wk 0), Post-Intervention (32-36 Wks), Follow-Up 1 (36-40 Wks), Follow-Up 2 (44-52 Wks), Follow-Up 3 (84-88 Wks)
  The investigators will examine whether sunburn occurrence decreased over time from pre- to post-intervention, specifically whether the odds of sunburn occurrence are lower for SHINE compared to standard education. An item from the Sun Habits Survey will ask students to report the number of sunburns they experienced within a specific time period.
  "In the past (time period), how many times did you have a red OR painful sunburn that lasted a day or more?" Minimum value = 0; Maximum value = 5 or more; Lower scores indicate a better outcome.
Change in Ultraviolet Radiation (UVR) Exposure Assessed Via UVR Monitor | Baseline (Wk 0), Post-Intervention (32-36 Wks), Follow-Up 1 (36-40 Wks), Follow-Up 2 (44-52 Wks), Follow-Up 3 (84-88 Wks)
  The investigators will examine whether UVR exposure decreased over time from pre- to post-intervention. 10% of all participants (evenly distributed across schools and conditions) will be asked to wear a UVR monitoring device immediately following each of the five assessments. The device will be used as an objective assessment of UVR exposure, and will provide information on the participant's UVR exposure over a seven day period.

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Wu, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT04341064/ICF_001.pdf